CLINICAL TRIAL: NCT03729700
Title: The Effect of Almonds on Facial Aesthetics and Modulation of the Microbiome and Lipidome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1257688
Record Dates: First submitted 2018-10-30; First posted 2018-11-05 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond supplementation (Experimental): The almond dose will be provided as 20% of total energy (20% E) in the diet. This dose was selected based on a previous randomized trial examining lipid parameters in response to 0, 10%, and 20% E as dietary almonds and a recent meta-analysis of intervention trials.
  Interventions: Other: Almond
- Control snack (No Intervention): The control snack will be a typical western diet snack. The calorie-matched control snack will be commercially available individually wrapped food products.

INTERVENTIONS:
Other: Almond — The almond dose will be provided as 20% of total energy (20% E) in the diet.
  Arms: Almond supplementation

SUMMARY:
The investigator hypothesizes that regular consumption of almonds will 1) improve the facial wrinkle severity in post-menopausal women, 2) improve the evenness of facial skin pigmentation, 3) diversify the gut microbiome and increase the short chain fatty acids in the blood, and 4) improve the skin barrier biophysical properties.

DETAILED DESCRIPTION:
This study will be a 24 week supplementation study that utilizes two study groups: 1) control group and 2) almond supplementation: 20% energy intake. This will be a randomized, rater-blinded, and controlled study. There will be a total of 60 subjects, with 30 assigned to the control group and 30 assigned to almond supplementation.

Subjects will be recruited from the UC Davis Dermatology Clinic, UC Davis Main campus, California State University- Sacramento, and from the surrounding community physicians and the community in a 100 mile radius. The greater Sacramento area has a population of over 2 million to draw from and recruitment will be conducted through the use of Social Media and flyer based recruitment. Postmenopausal women have previous been recruited successfully in a previous study. The study visits will be performed at the UC Davis Dermatology Clinic located at 3301 C Street, Suite 1400, Sacramento, CA 95816.

Investigators will collect medical history and current medications from study participants- this is outlined in the HIPAA form. The two intervention groups will consist of those receiving almonds and those that are receiving a calorie matched snack. The almond dose will be provided as 20% of total energy (20% E) in the diet. This dose was selected based on a previous randomized trial examining lipid parameters in response to 0, 10%, and 20% E as dietary almonds and a recent meta-analysis of intervention trials of tree nuts [5, 6]. The control snack will be a typical western diet snack (see Table 1) . The calorie matched snacks are commercially available prepackaged snack items that will be purchased from Costco. Once a subject has met inclusion criteria and has signed IRB consent, anthropometric data will be obtained, 1-24 hour recall will be collected, training will be provided for recording dietary records, and estimated caloric needs will be calculated. Estimated energy needs (EER) will be determined using the Mifflin-St. Jeor equation and total daily energy needs (TDE) calculated as EER x activity factor of 1.3-1.5 for sedentary to average activity, or a higher activity level as indicated. A representative example of a 60 year old woman, 5'4", 140 pounds with typical activity level yields TDE of approximately 1,600 - 1,800 kcal/day, and 20% E of 320-360 kcal/day. The intervention and control snacks would be 56.7 g of almonds and 56.7 g pretzel + one-24 g chewy granola bar, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Fitzpatrick skin types 1 and 2
* Able to follow dietary intervention and attend all study visits

Exclusion Criteria:

* Those with a nut allergy
* Current smokers, those that have smoked within the past year, and former smokers with greater than a 20 pack-year history of smoking, as smoking is a independent risk factor and serves as a confounder for the development of facial wrinkles
* Those with an autoimmune photosensitive condition or a known genetic condition with a deficiency in collagen production (such as Ehler-Danlos), as this can be a confounder for the development of facial wrinkles
* Those that already obtain 20% of their energy intake from nut consumption
* Those with implausible reported energy intakes of <1,000 kcal/d or >3,000 kcal/d
* Individuals who are unwilling to discontinue vitamin E containing supplements and food sources during the washout and intervention

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Post-menopausal women
Enrollment: 60 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Change in wrinkle severity | 24 weeks
  Photographs will be obtained at baseline, 8 weeks, 16 weeks, and 24 weeks. The images will be obtained with the 3D Clarity Pro® Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA) that has standardized positioning and lighting and iPad. The investigator has already validated this measurement tool against standard clinical grading of facial wrinkles.

SECONDARY OUTCOMES:
Change in facial pigmentation | 24 weeks
  Photographs will be obtained at baseline, 8 weeks, 16 weeks, and 24 weeks. The images will be obtained with the 3D Clarity Pro® Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA) that has standardized positioning and lighting and iPad. This system can assess facial pigmentation evenness and average intensity. The investigator has already validated this measurement tool against standard clinical grading of facial pigmentation.
Change in appearance of facial wrinkles on lateral canthi | 24 weeks
  Two blinded physician graders will grade the photographs obtained at each of the time points on the lateral canthi ("crow's feet").
Change in facial sebum production | 24 weeks
  Change in facial sebum production through the use of a Sebumeter, a commonly used device that measures sebum excretion rate. Sebum excretion rate will be measured at baseline, 8 weeks, 16 weeks, and 24 weeks.
Change in the serum profile | 24 weeks
  Change in the serum and sebum lipid profile for assessment of long chain/short chain fatty acid ratios and the NS ceramide content.
Change in sebum lipid profile | 24 weeks
  Change in the sebum lipid profile assessment of long chain/short chain fatty acid ratios and the NS ceramide content.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Department of Dermatology, Clinical Trials Unit, Sacramento, California, United States